CLINICAL TRIAL: NCT02017496
Title: Safety of Breast Conserving Treatment in Locally Advanced Breast Cancer Receiving Neoadjuvant Treatment
Acronym: NeoBCT
Status: Terminated | Type: Observational
Why Stopped: Too low inclusion rate
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Bjørn Naume, Principal investigator, Oslo University Hospital
Other Study IDs: S-08450d
Record Dates: First submitted 2013-10-23; First posted 2013-12-20 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer
Keywords: Breast cancer; locally advanced; neoadjuvant treatment; breast conserving surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sampling of primary tumor DNA and RNA is not included as a study specific procedure, but if the patient is included in a different ongoing protocol with tumor sampling, there is approval/allowance for using tumor tissue for the purpose of the current study (characteristics of the primary tumor that may predict residual tumor pattern and BCT success)
Oversight: Data Monitoring Committee: No

SUMMARY:
The study explores the safety of breast conserving treatment (BCT)(defined as complete removal of tumor deposits) after neoadjuvant treatment for locally advanced breast cancer.

DETAILED DESCRIPTION:
The standard breast surgical procedure of locally advanced breast cancer in Norway is mastectomy. There is increasing interest in performing breast conserving treatment (BCT) in locally advanced cases after chemotherapy or hormonal treatment - if there is a partial or complete clinical remission. To increase the evidence for the safety (no residual tumor) of such a procedure directly compared to mastectomy without compromising the safety of the treatment, a breast preserving procedure followed by an immediate mastectomy can be performed within a study. It would then be possible to study the margins after the breast preserving procedure as well as the tumor status in the rest of the breast.

Patients included in the study will receive neoadjuvant treatment followed by evaluation of the tumor reduction by magnetic resonance imaging (MRI) and selection of BCT candidates. Candidates will be prepared for BCT, and during the surgical procedure, BCT will be performed (as one surgical specimen) followed by immediate removal of the rest of the breast tissue (mastectomy). The BCT specimen and mastectomy specimen will be analysed for residual tumor cells. The tumor removal completeness of the BCT procedure can be evaluated, with comparison to the clinical and primary tumor characteristics, including analysis of the tumor biopsies and imaging before and during the neoadjuvant treatment, for selection of candidates for BCT in the future.

ELIGIBILITY:
Inclusion criteria:

* Patients with locally advanced breast cancer (cT3-4c, N0-3) with tumors > 5 cm, as determined by MRI, where the present guidelines include them for neoadjuvant systemic therapy
* Written informed consent (informed consent document to be approved by the Independent Ethics Committee) prior to study-related procedures and examinations.
* Female age > 18 years
* Able to comply with the protocol
* Histologically confirmed adenocarcinoma of the breast
* American Society of Anesthesiologist's physical status category 1 or 2 before surgery. Category 1 and 2 includes healthy patients and patients with only mild systemic disease, whereas category 3 includes patients with more serious systemic diseases (but still operable).

Exclusion criteria:

* Inflammatory breast cancer or diffuse locoregional involvement of the skin
* Stage IV - metastatic disease
* Locoregional relapse of earlier breast cancer
* Inability (irrespective of reason) to receive the recommended neoadjuvant treatment, - as decided by the treating physician.
* American Society of Anesthesiologist's physical status category 4-5

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to neoadjuvant treatment at the University Hospitals in Norway who are candidates for neoadjuvant treatment.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
1 The presence of viable tumor cells at the margins and in the mastectomy specimen after conducted breast preserving resection followed by mastectomy in the same procedure | 24 weeks after start of neoadjuvant treatment (at surgery)
  The surgical specimens will be analysed after surgery, and the results of these analyses will be the basis for the final end point measurements.

SECONDARY OUTCOMES:
Tumor molecular marker characteristics related to complete resection by BCT | 24 weeks after start of neoadjuvant treatment (at surgery)
  Tumor molecular marker characteristics, MRI, mammography (Mx) and ultrasound (US) results and clinical parameters in patients with residual tumor cells in the mastectomy specimen compared to those with no tumor cells

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Naume, Professor, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway